CLINICAL TRIAL: NCT05062655
Title: Nterest of Drug Reconciliation to Ensure the Continuity of the Treatment at Discharge
Brief Title: Interest of Drug Reconciliation to Ensure the Continuity of the Treatment at Discharge
Acronym: ICOCON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHM-2021/S21/09
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-09

CONDITIONS: Hospitalized Patient
Keywords: Medication reconciliation; Continuity; Town-hospital network

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug reconciliation (Experimental): Drug reconciliation and transmission to pharmacist
  Interventions: Other: Drug reconciliation
- standard (No Intervention)

INTERVENTIONS:
Other: Drug reconciliation — Drug reconciliation information transmission to pharmacist interview with the patient
  Arms: Drug reconciliation

SUMMARY:
From a regulatory point of view, medication reconciliation is a necessary process to ensure safe medication management for patients. According to national studies and the international scientific literature, the information received by patients and health professionals at discharge from hospital is insufficient.

Medication reconciliation at discharge reduces medication errors and rehospitalisation, but few studies have been conducted on the impact of a coordinated and reliable care pathway on medication continuity.

The iCoCon study will enable a new healthcare organisation to be set up in order to improve the quality of the patient pathway and the patient's medication management.

This new organisation is part of the policy of continuous improvement of the quality and safety of care

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patient
* Patient with a drug treatment with a particular mode of supply
* Paediatric patient or an adult patient.
* First inpatient stay over the inclusion period from late 2021 to late 2022

Exclusion Criteria:

* Patient under curatorship or guardianship
* Patient residing abroad
* No free, informed and written consent obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-08 (Estimated); Study Completion 2022-12-08 (Estimated)

PRIMARY OUTCOMES:
Value of a coordinated and reliable pathway when patients are discharged from the institution via drug reconciliation to ensure the continuity of patients' treatment | 1 month after inclusion
  Value of coordinated pathway is evaluated by number of days of treatment interruption between patient discharge and provision of treatment to the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France